CLINICAL TRIAL: NCT06967519
Title: OPTImizing Malaria And HIV Treatment in a Shifting Landscape in Africa
Acronym: OPTIMAH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000039347; 2R01HD068174-11A1 (NIH)
Record Dates: First submitted 2025-04-23; First posted 2025-05-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Malaria; Hiv
MeSH Terms: conditions — Malaria; Acquired Immunodeficiency Syndrome | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: Only Busia participants (HIV-infected and HIV-uninfected, Cohorts 3 and 4) will be enrolled and then randomized to receive either artemether- lumefantrine (AL) or artesunate-amodiaquine (AS-AQ) for each episode of malaria which occurs over longitudinal follow-up in year one. During year 1, they will continue to receive the same antimalarial each time they are treated for uncomplicated malaria. In year two, those randomized to the AL arm will begin to receive an alternating regimen for each subsequent malaria episode (AS-AQ, then AL, then AS-AQ, etc..). CLHIV, ages 5-17 years, will be identified from respective registers at Baylor-Uganda (in Kampala) and the Masafu HIV clinic (and nearby clinics) in Busia Uganda. HIV-uninfected children, also ages 5-17 years, will be enrolled from catchment areas at these two sites. Recruitment will be balanced by age and sex.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CLHIV on DTG- Kampala (Cohort 1) (Experimental): CLHIV on DTG living in the low transmission malaria setting of Kampala
  Interventions: Drug: Artemether-lumefantrine (AL); Drug: artesunate-amodiaquine (AS-AQ)
- HIV-uninfected children- Kampala (Cohort 2) (No Intervention): HIV-uninfected children living in the low malaria transmission site of Kampala (control)
- CLHIV on DTG- Busia (Cohort 3) (Experimental): CLHIV on DTG living in the high malaria transmission site of Busia
  Interventions: Drug: Artemether-lumefantrine (AL); Drug: artesunate-amodiaquine (AS-AQ)
- HIV-uninfected children- Busia (Cohort 4) (No Intervention): HIV-uninfected children living in high malaria transmission site of Busia (control)

INTERVENTIONS:
Drug: Artemether-lumefantrine (AL) — Participants will receive the dispersible formulation of AL with contains 20 mg artemether, 120 mg of lumefantrine
  Arms: CLHIV on DTG- Busia (Cohort 3); CLHIV on DTG- Kampala (Cohort 1)
Drug: artesunate-amodiaquine (AS-AQ) — Children will receive the tablet formulations of Artesunate Amodiaquine using weight based dosing
  Arms: CLHIV on DTG- Busia (Cohort 3); CLHIV on DTG- Kampala (Cohort 1)

SUMMARY:
A longitudinal study with four parallel cohorts with each participant followed for 2 years: two cohorts in Busia (high malaria transmission site) and two cohorts in Kampala (low malaria transmission). Each site will have a cohort of children living with HIV (CLHIV) and HIV- uninfected children and will be age-matched, enrolled in parallel, and followed for two years. All children will be enrolled without malaria infection, as determined by a negative blood smear at baseline.

DETAILED DESCRIPTION:
CLHIV will be maintained on a dolutegravir (DTG) based regimen for >2 weeks prior to enrolment to ensure steady state. All children in Busia (HIV-infected and HIV-uninfected) will be enrolled and then randomized to receive either artemether- lumefantrine (AL) or artesunate-amodiaquine (AS-AQ) for each episode of malaria which occurs over longitudinal follow-up in year one. During year 1, they will continue to receive the same antimalarial each time they are treated for uncomplicated malaria. In year two, those children randomized to the AL arm will begin to receive an alternating regimen for each subsequent malaria episode (AS-AQ, then AL, then AS-AQ, etc..). If local/national guidelines in Uganda for malaria change during the course of the study, the treatment arms will be altered as applicable. Aim 1: To what extent does DTG impact, BMI, body composition and metabolic changes? Aims 2 and 3: Are there critical drug-drug interactions between DTG and first line artemisinin-based combination therapies (ACTs)? Do these changes impact HIV and malaria outcomes? What is the status of ACT resistance and its relationship to PK exposure?

MALARIA CASE DEFINITION:

Uncomplicated malaria (all of the following)

* Fever (≥ 37.5ºC axillary) or history of fever in the previous 24 hours
* Positive thick blood smear (any parasitemia)
* Absence of severe malaria Severe malaria
* Evidence of severe malaria as per WHO criteria

ELIGIBILITY:
Inclusion Criteria:

* Agreement to come to the clinic for all follow-up evaluations
* Provision of informed consent and assent (as appropriate)
* Residency within approximately 30 km of the study clinic
* Negative blood smear for malaria (all sites)
* For Children and adolescents living with HIV

  * Confirmed HIV infection
  * On DTG-based regimen for ≥14 days
* For HIV-uninfected children - documentation of HIV-negative status by at least 1 assay

Exclusion Criteria:

* Significant comorbidities such as malignancy, active TB, chronic/active hepatitis B/C, diabetes, severe acute malnutrition, mitochondrial disorders
* Receipt of known CYP interacting drugs at enrolment (except HAART) - see list of disallowed medications
* Anemia defined by hemocue (Hb < 7.0) at the time of enrolment
* Signs of uncomplicated or severe malaria at the time of enrollment
* Prior intolerance to AL or AS-AQ (for those in Busia only)
* Pregnancy at enrolment (testing done at enrollment for all those of child-bearing age)
* Concurrent enrolment in another research study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | baseline and 2 years
  Change in BMI from baseline and 2 years in kg/m² (Cohort 1 + 3 vs Cohort 2 + 4)
Drug pharmacokinetic (PK) exposure | baseline up to 2 years
  Comparison of drug exposure by DTG and anti-malarial regimen using Area under the curve (AUC) (Cohort 1 vs 3)
Drug pharmacokinetic exposure | baseline up to 2 years
  Comparison of drug exposure by DTG and anti-malarial regimen using Area under the curve (AUC) (Cohort 3 vs 4)
Recurrence rate of malaria | 28 days and 42 days
  To assess the 28 and 42 day efficacy of AL and AS-AQ for the treatment of uncomplicated malaria in children with and without HIV.

SECONDARY OUTCOMES:
Average change in glucose sensor readings | every 6 months up to 2 years
  Change in average of continuous glucose monitor readings over the last 10 days. (Cohorts 1 vs 2)
Change in insulin resistance (HOMA-IR) | baseline and 2 years
  Change in HOMA-IR in those living with and without HIV. (Cohorts 1+3 vs 2+4)
Change in Body Mass Index (BMI) | baseline and 2 years
  Change in BMI in children living with HIV from baseline and 2 years in kg/m² (Cohort 1 vs 3)
Pharmacokinetic parameters | immediately post drug exposure (Day 1)
  AUC (0-8h) and AUC (last) for lumefantrine and DEAQ. (Cohorts 1 and 3)
Change in HIV viral load | every 6 months up to 2 years
  Change of HIV viral load suppression in those on DTG vs children not living with HIV. (Cohorts 1 vs 3)
Malaria treatment outcome | 28 days and 42 days
  28 and 42 day antimalarial treatment efficacy in those on DTG vs Children not living with HIV, as measured by peripheral blood smears
HIV genotypic resistance to DTG | baseline and 2 years
  Resistance to DTG (binary measures as yes/no) as measured by HIV molecular genotype (Cohort 1 and 3)
Artemisinin PK concentration-time profile | During treatment of malaria episodes over 2 years
  Area under the plasma concentration versus time curve (AUC) in those receiving AL vs AS-AQ. (Cohorts 3 and 4)
Rate of parasite clearance | During treatment of malaria episodes over 2 years
  Parasite clearance half-life in those treated with AL vs AS-AQ. (Cohorts 3 and 4)
Rate of parasite clearance and HIV | During treatment of malaria episodes over 2 years
  Parasite clearance half-life in those living with HIV and those not living with HIV. (Cohorts 3 and 4)
Gametocyte quantity | At the time of presentation with malaria up to 2 years
  Quantity of gametocytes in the peripheral blood in those treated artemisinin sensitive vs resistant infections. (Cohorts 3 and 4)

OTHER OUTCOMES:
Time to resistance | up to 2 years
  Time to resistance mutation in days. (Cohort 3 and 4)
K13 mutations | up to 2 years
  Rate of K13 mutation and Artemisinin partial resistance. (Cohort 3 and 4)
Prevalence of mutations in malaria transporters | During treatment of malaria episodes over 2 years
  Change in mutation prevalence of pfcrt and pfmdr1 in those treated with AL vs AS-AQ for malaria.(Cohort 3 and 4)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Parikh, M.D., MPH, Principal Investigator — Yale School of Public Health
Locations (2):
- Uganda (2):
  - Baylor- Uganda, Kampala
  - Infectious Disease Research Collaboration (IDRC), Kampala

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified, and shared on clinepidb.org upon conclusion of the study